CLINICAL TRIAL: NCT06431334
Title: Protein Requirements Amongst Male Masters-Level Athletes Following a Cycling Exercise Bout as Determined by the Indicator Amino Acid Oxidation Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A06-M25-23A
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Increased Metabolic Requirements; Dietary Reference Intakes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Masters Level Cyclists (Experimental): Participants are to be randomly assigned varying levels of amino acid intakes ranging between 0.2 to 2.8 g/kg/d
  Interventions: Dietary Supplement: Amino Acid Intake

INTERVENTIONS:
Dietary Supplement: Amino Acid Intake — Amino acid intakes will vary between 0.2 to 2.8 g/kg/d

SUMMARY:
Masters level cyclists are a population above the age of 35 years who frequently participate in prolonged as well as heavy-volume training. Like most endurance-trained athletes, a greater recommended dietary allowance (RDA) for protein of 1.2-1.4 g/kg/bw is suggested.

Dietary protein intake is vital for maximizing the benefits of training and ensuring optimal recovery. Dietary recommendations traditionally have been determined through nitrogen balance techniques, however, recent research indicates how this method is potentially underestimating protein requirements. Therefore, there is a need to reassess current dietary recommendations in order to meet the demands of physical activity for highly active populations.

Recent efforts to understand protein requirements during rest and following exercise have been completed using the indicator amino acid technique (IAAO). This non-invasive method is reported to provide a robust measure of protein requirements. However, there is limited work in older (≥60 years) active populations.

The purpose of this study is to measure the protein requirements in master cyclists, following an endurance training session, using the non-invasive IAAO technique.

ELIGIBILITY:
Inclusion Criteria:

* 18.5< BMI <35 kg/m^2
* Overtly healthy masters level cyclists ≥65 years
* Masters level cyclist training (>4 days per week; ~100 km per week)
* Body mass stable over previous 6-months
* Availability for multiple metabolic trials (~7 trials)
* Ability to travel to and from laboratory facility

Exclusion Criteria:

* Recent history of weight loss or weight gain (>5% body weight)
* Uncontrolled hypertension
* ≥2 chronic diseases (e.g. diabetes, osteoporosis, dyslipidemia)
* Acute illness that could affect protein metabolism (HIV, renal dysfunction, influenza)
* Currently using anti-inflammatory medications
* Inability to adhere to study protocol (i.e., alcohol, caffeine, dietary restrictions)
* Regular tobacco user
* Illicit drug use
* Habitually ingesting ≥3 g/kg/bw

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
13CO2 Excretion | 7-weeks
  Measured by continuous-flow isotope ratio mass spectrometry

SECONDARY OUTCOMES:
L[13C]phenylalanine Oxidation | 7-weeks
  Measured by gas chromatography-mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada